CLINICAL TRIAL: NCT01519635
Title: Effect of Aliskiren 300mg and Hydrochlorothiazide 25mg on Kidney Oxygenation in Patients With Stage 1 and 2 Hypertension: a BOLD-MRI Study
Brief Title: Effect of Aliskiren and Hydrochlorothiazide on Kidney Oxygenation in Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Michel Burnier, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011DR3137
Record Dates: First submitted 2012-01-06; First posted 2012-01-27 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Kidney oxygenation; Stage 1 or 2 hypertension; BOLD-IRM
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Active Comparator): Aliskiren 150 to 300 mg once a Week for 8 weeks
  Interventions: Drug: Aliskiren
- Hydrochlorothiazide (Active Comparator): HCTZ 12.5 - 25 mg/d once a day for 8 weeks
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Aliskiren — Drug therapy will be started with an initial 2 weeks on Aliskiren 150 mg followed by a titration to 300 mg Aliskiren if the treatment is well tolerated. A first baseline measurements will be performed before initiating therapy and a second after 8 weeks of treatment (24h after last drug intake) to assess the chronic effect.
  Other Names: Rasilez
  Arms: Aliskiren
Drug: Hydrochlorothiazide — Drug therapy will be started with an initial 2 weeks HCTZ 12.5 mg followed by a titration to 25 mg HCTZ if the treatment is well tolerated. A first baseline measurements will be performed before initiating therapy and a second after 8 weeks of treatment (24h after last drug intake) to assess the chronic effect.
  Other Names: Esidrex
  Arms: Hydrochlorothiazide

SUMMARY:
The goal of this project is to evaluate the chronic effect (8 weeks) of RASILEZ 300mg (aliskiren) on renal tissue oxygenation in patients with stage 1-2 hypertension, and to compare the chronic effect (8 weeks) of RASILEZ 300mg (aliskiren) on renal tissue oxygenation in patients with stage 1-2 hypertension with these effects with those of ESIDREX 25mg (hydrochlorothiazide).

DETAILED DESCRIPTION:
36 patients with arterial hypertension stage 1-2 (blood pressure: 140/90 and 180/110 mm Hg) will be included in this study and randomized to two groups of 18 patients each: one group will receive RASILEZ 300mg (aliskiren) and one group ESIDREX 25mg (hydrochlorothiazide).

After a two week washout of antihypertensive drugs, baseline and the chronic effect (8 week study drug) of each group will be studied with precise renal hemodynamic measurements (inulin clearance, PAH renal plasma and blood flow, sodium and endogenous lithium excretion, plasma renin, plasma aldosterone, urinary sodium and potassium) and assessment of renal oxygenation with BOLD-MRI (blood oxygen level detection - magnetic resonance imaging).

Drug therapy will be started with an initial 2 weeks on Rasilez 150 mg or HCTZ 12.5 mg followed by a titration to 300 mg Rasilez and 25 mg HCTZ if the treatment is well tolerated. In both groups: a first baseline measurements will be performed before initiating therapy and a second after 8 weeks of treatment (24h after last drug intake) to assess the chronic effect.

Patients already on treatment with antihypertensive drugs can be included in this study, but will undergo a 'wash-out' period of two weeks. After obtaining informed consent, baseline physical examination and office blood pressure measurement will be performed. Office blood pressure will be measured according to the guidelines of the European Society on Hypertension and European Society of Cardiology (ESH-ESC practice guidelines) by an experienced physician. Moreover, patients will measure their home blood pressure twice daily: after 5 minutes of sitting quietly, three measures spaced by 1-2 minutes will be taken in the morning and in the evening. For this purpose, an Omron 705 IT device will be provided to the participants; this device has been widely tested in clinical practice and has been validated for use in clinical studies (12).

Throughout the study, the participants will continue his/her regular diet. The goal should be to keep the salt intake as stable as possible during the study, since salt intake alters the R2* signal. Salt intake will be verified each time before BOLD-MRI measurement by a 24h urine collection (dosing volume, creatinine- and sodium-concentration).

To complete the study we decid to test the acute effect of aliskiren 300mg and Esidrex (hydrochlorthiazide) 25mg in 6 healthy volunteers. We will measure the cortical and medullary R2* signal before drug intake and 3 hours after drug administration. Each participant will take the two drugs in a randomised crossover design. A wash-out period of two week between the two administration will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Tolerance to study drugs
* Age > 18 years
* Arteria hypertension stage 1-2 (blood pressure: 140/90 and 180/110 mm Hg)
* Normal renal function
* Availability to give informed consent

Exclusion Criteria:

* Intolerance to study drugs
* Renal artery stenosis
* Hyperkalaemia > 5.0 mmol/l
* Contra-indications to the use of PAH, inulin or Lithium
* Asthma
* Pychiatric illness
* No estimated easy vascular venous access for placement of two peripherical venous catheters in forearms
* Contra-indication to MRI-imaging: Claustrophobia or Pacemaker or other implanted metal device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Burnier, Professor, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Pruijm M, Hofmann L, Maillard M, Tremblay S, Glatz N, Wuerzner G, Burnier M, Vogt B. Effect of sodium loading/depletion on renal oxygenation in young normotensive and hypertensive men. Hypertension. 2010 May;55(5):1116-22. doi: 10.1161/HYPERTENSIONAHA.109.149682. Epub 2010 Mar 22. PMID 20308608
- [Result] Vakilzadeh N, Muller ME, Forni V, Milani B, Hoffman L, Piskunowicz M, Maillard M, Zweiacker C, Pruijm M, Burnier M. Comparative Effect of a Renin Inhibitor and a Thiazide Diuretic on Renal Tissue Oxygenation in Hypertensive Patients. Kidney Blood Press Res. 2015;40(5):542-54. doi: 10.1159/000368530. Epub 2015 Oct 26. PMID 26501147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 patients were screened in a single centre (service of Nephrology, CHUV, Lausanne)
Pre-assignment Details: 24 patients were enrolled but 4 were excluded because of the lack of adequate venous access or for other reasons.
Groups:
- Aliskiren: Aliskiren: Drug therapy will be started with an initial 2 weeks on Aliskiren 150 mg followed by a titration to 300 mg Aliskiren if the treatment is well tolerated. A first baseline measurements will be performed before initiating therapy and a second after 8 weeks of treatment (24h after last drug intake) to assess the chronic effect.
  11 patients were enrolled and completed the study
- Hydrochlorothiazide: Hydrochlorothiazide: Drug therapy will be started with an initial 2 weeks HCTZ 12.5 mg followed by a titration to 25 mg HCTZ if the treatment is well tolerated. A first baseline measurements will be performed before initiating therapy and a second after 8 weeks of treatment (24h after last drug intake) to assess the chronic effect.
  Finally 9 patients were enrolled and completed the study
Period: Overall Study
Arm/Group | Aliskiren | Hydrochlorothiazide
Started | 12 | 12
Completed | 11 | 9
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — No possibility to put a catheter | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Aliskiren: Patients with essential hypertension stage 1 and 2 .
- HCTZ: Patients with essential hypertension stage 1 and 2
- Total: Total of all reporting groups
Arm/Group | Aliskiren | HCTZ | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (8.6) | 49.7 (15) | 52.7 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Switzerland | 11 | 9 | 20
blood pressure [Mean (Standard Deviation); unit: mmHg] | 150 (10.7) | 141 (12.9) | 146 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Renal Oxygenation Changes After Chronic Treatment With Aliskiren or Hydrochlorothiazide
Description: Changes in R2* at between week 0 and week 8 as measured by BOLD MRI in the cortex and medulla of the kidney
Time Frame: week 0 vs week 8
Measure: Mean (Standard Error); unit: 1/sec
Arm/Group | Aliskiren | Hydrochlorothiazide
Number analyzed (Participants) | 11 | 9
1/sec
  Cortex week 0 | 20.5 (1) | 19.5 (1)
  Cortex week 8 | 19.5 (1) | 20.5 (1)

ADVERSE EVENTS:
Groups:
- Aliskiren: Aliskiren: Drug therapy has been started with an initial 2 weeks on Aliskiren 150 mg followed by a titration to 300 mg Aliskiren if the treatment is well tolerated. A first baseline measurements will be performed before initiating therapy and a second after 8 weeks of treatment (24h after last drug intake) to assess the chronic effect.
- Hydrochlorothiazide: Hydrochlorothiazide: Drug therapy has been started with an initial 2 weeks HCTZ 12.5 mg followed by a titration to 25 mg HCTZ if the treatment is well tolerated. A first baseline measurements will be performed before initiating therapy and a second after 8 weeks of treatment (24h after last drug intake) to assess the chronic effect.
  No side effect were observed and all patients finished the sudy in this treatment arm
Arm/Group | Aliskiren | Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
Small number of patients who completed the study. Overall underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No